CLINICAL TRIAL: NCT06596135
Title: Open-Label Extension Study of Setmelanotide in Patients With a Rare Genetic, Syndromic or Acquired Disease of the MC4R Pathway
Brief Title: Open-Label Extension Study of Setmelanotide
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RM-493-042
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Obesity Associated With Defects in Leptin-melanocortin Pathway
Keywords: setmelanotide; RM-493; obesity; melanocortin 4 receptor; hypothalamic obesity
MeSH Terms: conditions — Obesity; Sexual Infantilism | interventions — setmelanotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Setelanotide (Open-label) (Experimental): Once daily (QD) subcutaneous injection of setmelanotide
  Interventions: Drug: Setmelanotide

INTERVENTIONS:
Drug: Setmelanotide — Open-label daily injections of setmelanotide
  Other Names: RM-493; Imcivree

SUMMARY:
This is an open-label extension study designed to evaluate the long-term safety and tolerability of continued setmelanotide treatment in male and female patients ≥2 years of age who have completed or transitioned from a previous study with setmelanotide for rare genetic, syndromic, or acquired diseases of obesity upstream of the MC4R pathway.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and females ≥2 years of age who have completed a previous setmelanotide clinical study and who have a condition or indication for which Rhythm plans further clinical development.
* Agree to use a highly effective form of contraception and follow the study contraception requirements throughout study duration and for 90 days after.
* Demonstrated clinical benefit in the previous setmelanotide study, as determined by the Investigator.

Key Exclusion Criteria:

* Any gene variant, syndromic, or acquired disease for which setmelanotide is currently approved in the United States (i.e., patients eligible for commercial setmelanotide (IMCIVREE®).
* Any new or worsening depression resulting in suicidal thoughts and/or behaviors.
* Discontinuation from a previous setmelanotide study.
* History or close family history (parents or siblings) of melanoma.
* Pregnant and/or breastfeeding women

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of setmelanotide assessed by frequency and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, MD, Study Chair — Rhythm Pharmaceuticals, Inc.
Locations (13):
- United States (13):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - UC San Diego- Rady Children's Hospital, San Diego, California
  - University of Florida at Gainesville, Gainesville, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Children's Minnesota, Saint Paul, Minnesota
  - University of Buffalo, Getzville, New York
  - M3 Wake Research, Inc, Raleigh, North Carolina
  - Geisinger Health System, Danville, Pennsylvania
  - WR-ClinSearch, Chattanooga, Tennessee
  - Vanderbilt University School of Medicine, Nashville, Tennessee
  - Seattle Children's Research Institute, Seattle, Washington
  - Marshfield Clinical Research Institute, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: No